CLINICAL TRIAL: NCT00259402
Title: Phase II Open-label Single Arm Study of Oxaliplatin Combined With Cisplatin and 5FU in Advanced Esophagus Cancer Patients
Brief Title: Oxaliplatin in Esophagus Cancer (Advanced) 1st Line
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC_7127
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; Cisplatin; Fluorouracil

ARMS (1):
- Oxaliplatin (Experimental)
  Interventions: Drug: Oxaliplatin + cisplatin + 5-Fluorouracil (5-FU)

INTERVENTIONS:
Drug: Oxaliplatin + cisplatin + 5-Fluorouracil (5-FU) — OXALIPLATIN 60 mg/m2/d, CISPLATIN 55 mg/m2/d, 5-FU 600 mg/m2/d with dose range and followed by radiotherapy

SUMMARY:
* To determine the activity and efficacy of the schema specified as dose regimen
* To determine the safety and tolerability of the oxaliplatin-cisplatin and 5FU

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* Patients with histologically proven epidermoid carcinoma or adenocarcinoma of esophagus or stomach, with unresectable or metastatic disease;
* No previous treatment with chemotherapy or radiotherapy
* Measurable lesion (uni or bidimensional)

Exclusion Criteria:

* Creatinin clearance <50 mL/min
* Total bilirubin >1.5*ULN (Upper Limit of Normal)
* AST/ALT > 2.5*ULN
* Total White Blood Cell <1.500.000/mL
* Platelet count <100.000.000/mL
* symptomatic sensitive peripheral neuropathy
* pregnant or breast-feeding women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2000-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoints include tumor response, progression free and overall survival. | Throughout the whole study

SECONDARY OUTCOMES:
Safety endpoints include summary of adverse events assessed by history, physical exams and laboratory evaluations. | Throughout the whole study duration

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Barcelona, Spain